CLINICAL TRIAL: NCT05773612
Title: Rock Steady Boxing: A Community Based In Person Class for Patients With Parkinson Disease
Brief Title: Rock Steady Boxing: A Community Based In Person Class
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of St. Augustine for Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-0401-498
Record Dates: First submitted 2022-10-22; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rock Steady Boxing classes (Other): The Rock Steady Boxing classes are 60-90 minutes in duration twice a week and include the following 4 components: (1) active warm up (2) functional mobility exercises (3) whole body strengthening exercises and (4) non-contact boxing exercises.
  Interventions: Other: Rock Steady Boxing Class

INTERVENTIONS:
Other: Rock Steady Boxing Class — Rock Steady Boxing is a non-contact fitness program designed specifically for people with Parkinson's Disease.

SUMMARY:
The purpose of this study is to evaluate the feasibility and effectiveness of a non-contact Rock Steady Boxing class delivered to participants with Parkinson's Disease via an in-person community-based program. The study will also assess the overall feasibility of integrating an in-person community program within a neuromuscular course in a Doctor of Physical Therapy program.

Specific Aim: To examine the effects of an in-person community-based Rock Steady Boxing class on the functional mobility, functional endurance, cardiovascular capacity, visual-motor reaction times, quality of life, mood/affect and overall physical activity completion and fear of falling on individuals with Parkinson's Disease.

DETAILED DESCRIPTION:
Participants will be recruited directly from the the Brain Center (non-for-profit neurology clinic). Participants will be educated on the study but advised that their participation is voluntary and researchers will not coerce boxers to participate in the study. Once a participant agrees to participate, the Informed consent will be completed. During this time, participants will be told their participation is voluntary and they can quit at any time. he primary interventions being assessed in this study include the in-person Rock Steady Boxing Class offered at USAHS once per week. Prior to attending the Rock Steady Boxing classes, all participants must be provided with medical clearance from a referring medical doctor. The Rock Steady Boxing classes are 60-90 minutes in duration and include the following 4 components: (1) active warm up (2) functional mobility exercises (3) whole body strengthening exercises and (4) non-contact boxing exercises. During the classes, boxers' vitals are assessed using health rate monitors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age Range: 18 years or older
3. History of Parkinson's Disease between Hoehn and Yarh stages I and IV
4. Medical clearance from a referring medical doctor
5. Able to complete all assessments
6. Willing to complete a weekly exercise log

Exclusion Criteria:

1. Unable to complete the assessments.
2. Pregnant or is expected to become pregnant during study
3. Other reasons that may limit participation in exercises. -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-07 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes over time in Activities-Specific Balance Confidence Scale (ABC) from baseline to one year | Baseline, 3 months, 6-months and 1-year post intervention
  The ABC is a self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness.
Changes in Falls Efficacy Scale - International from baseline to 1-year post | Baseline, 3 months, 6-months and 1-year post intervention
  A self-administered questionnaire designed to assess fear of falling in mainly community-dwelling older population
Changes in Parkinson's Disease Fatigue Scale from baseline to 1-year post | Baseline, 3 months, 6-months and 1-year post intervention
  A patient-rated scale that measures fatigue
Changes in Parkinson's Disease Questionnaire -39 from baseline to 1-year post | Baseline, 3 months, 6-months and 1-year post intervention
  A 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month.
Changes in Physical Activity Scale for the Elderly (PASE) from baseline to 1-year post | Baseline, 3 months, 6-months and 1-year post intervention
  The PASE measures the level of self-reported physical activity in individuals aged 65 years old or older and is comprised of items regarding occupational, household, and leisure activity during the previous 7-day period.
Changes in Berg Balance Test from baseline to 1-year post | Baseline, 3 months, 6-months and 1-year post intervention
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks.
Changes in 10-Meter Walk Test from baseline to 1-year post | Baseline, 3 months, 6-months and 1-year post intervention
  The 10 Meter Walk Test is a performance measure used to assess walking speed in meters per second over a short distance.
Changes in 6-Minute Walk Test from baseline to 1-year post | Baseline, 3 months, 6-months and 1-year post intervention
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance.
Changes in Time Up and Go (TUG) from baseline to 1-year post | Baseline, 3 months, 6-months and 1-year post intervention
  Measure of function with correlates to balance and fall risk
Changes in Self-Efficacy for Exercise from baseline to 1-year post | Baseline, 3 months, 6-months and 1-year post intervention
  Self report measure of exercise self-efficacy
Changes in Anticipatory & Compensatory Postural Assessment form baseline to 1-year post | Baseline, 3 months, 6-months and 1-year post intervention
  Electromyography measure of postural stability in standing
Changes in Rock Steady Boxing Questionnaire from 3-month post to 1-year post intervention | 3 months, 6-months and 1-year post intervention
  Self assessment of mobility and quality of life
Changes Physical Activity Intensity Monitoring from baseline to 1-year post intervention | Baseline, 3 months, 6-months and 1-year post intervention
  Heart rate monitoring during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Garcia, EdD, Principal Investigator — University of St Augustine for Health Science
Locations (1):
- University of St Augustine for Health Science, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in rehabilitation for individuals with Parkinson's Disease. Data or samples shared will be coded, with no Private Health Information included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial Individual Patient Data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement.